CLINICAL TRIAL: NCT05909046
Title: A Randomized Controlled Trial of Diabetes Screening Immediately Postpartum (DIP) - Follow up Study: Patient Perspectives on Postpartum Interventions to Improve Future Maternal CARdiovascular hEalth After Gestational Diabetes (PP CARE)
Brief Title: A Randomized Controlled Trial of Diabetes Screening Immediately Postpartum (DIP) and Follow Up PP CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kartik K Venkatesh, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023H0189
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pre-Gestational Diabetes; Type2diabetes; Pregnancy in Diabetic; Pregnancy, High Risk; Gestational Diabetes; Gestational Diabetes Mellitus in the Puerperium
Keywords: 2-hour oral glucose tolerance test (OGTT); Pregnancy; diabetes mellitus screening; postpartum; cardiometabolic health; cardiovascular health; type 2 diabetes; prediabetes
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes, Gestational; Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate inpatient postpartum OGTT (Active Comparator): The intervention includes immediate inpatient postpartum 2-hour oral glucose tolerance test (OGTT) prior to delivery discharge
  Interventions: Diagnostic Test: Immediate inpatient postpartum OGTT
- Standard of care (Other): Standard of care is 4-12 week outpatient postpartum OGTT
  Interventions: Diagnostic Test: Standard of care 4-12 week postpartum OGTT

INTERVENTIONS:
Diagnostic Test: Immediate inpatient postpartum OGTT — The intervention includes immediate inpatient postpartum 2-hour oral glucose tolerance test (OGTT) prior to delivery discharge
  Arms: Immediate inpatient postpartum OGTT
Diagnostic Test: Standard of care 4-12 week postpartum OGTT — Standard of care is 4-12 week outpatient postpartum OGTT
  Arms: Standard of care

SUMMARY:
DIP : To conduct a pragmatic, non-blinded randomized controlled trial (pRCT) of immediate in-patient postpartum OGTT prior to delivery discharge (intervention) versus 4-12 week outpatient postpartum OGTT (current standard care) to improve the frequency of post-partum diabetes screening among individuals with a pregnancy complicated by GDM.

Follow up PP CARE: To engage with individuals with a history of GDM through a patient-centered mixed-methods survey and qualitative assessment to evaluate the barriers to and facilitators of Cardiovascular health (CVH) counseling and risk-reduction postpartum at the patient and healthcare system levels inclusive of Social determinants of health (SDOH) and structural factors, as well as patient preferences and perspectives on CVH and wellness interventions

DETAILED DESCRIPTION:
DIP: Individuals with gestational diabetes (GDM) during pregnancy have up to a 10-fold increased risk of developing of T2DM. Postpartum screening facilitates detection of impaired glucose tolerance and diabetes mellitus with the possibility for subsequent preventive and treatment interventions. The American College of Obstetricians and Gynecologists (ACOG) and the American Diabetes Association (ADA) recommend screening individuals with GDM postpartum with a 75-g, 2-hour oral glucose tolerance test (OGTT) that includes a fasting blood glu-cose.4,6 This is historically performed at 4-12 weeks so that it will coincide with the timing of the typical postpartum visit. However, the rate of postpartum screening with the recommended method are low, as many individuals do not seek timely postpartum care-only a quarter to one half of individuals undergo diabetes screening in the first year postpartum. Multiple structural barriers exist for patients and healthcare providers to effectively complete postpartum diabetes screening via the current recommended method. An immediate postpartum OGTT has been proposed as an alternative to the current standard practice which is generally performed between 4-12 week postpartum OGTT at the routine postpartum visit. An immediate OGTT has comparable performance characteristics for detection of impaired glucose tolerance and diabetes compared with a 4-12 week postpartum OGTT.

Follow up PP CARE: Postpartum adverse CVH is a critical public health problem and contributes to persistent and inequitable maternal health. Adverse cardiovascular health outcomes after delivery, including hypertension, dyslipidemia, diabetes, and obesity, are frequent and a major source of maternal morbidity and mortality. Ultimately, these conditions increase the risk of long-term cardiovascular disease which affects 60 million women in the United States (US). It represents the leading cause of death, contributing to 1 in 5 deaths in women in the US. Despite these epidemiologic associations, relatively less research exists on prevention, recognition and treatment of adverse CVH in high-risk postpartum women before the occurrence of clinical disease. Further, adverse CVH is more common among individuals who experience an adverse pregnancy outcome (APO), as well as adverse social determinants of health (SDOH), including self-identified minoritized race or ethnicity as a proxy for racism, low socioeconomic status, housing and food insecurity, and limited access to healthcare.

ELIGIBILITY:
DIP - Inclusion Criteria:

* Immediately postpartum individuals during their delivery hospital admission
* ≥ 18 years old with the ability to give informed consent.
* Diagnosed with GDM during pregnancy by:

  * Elevated one-hour 50-gram glucose challenge test any time during pregnancy AND provider documentation of gestational diabetes (NOT pregestational diabetes) diagnosis OR
  * Two elevated values on a 3-hour 100-gram glucose tolerance test any time in pregnancy AND provider documentation of gestational diabetes (NOT pregestational diabetes) diagnosis
* English or Spanish speaking
* Receiving prenatal and postpartum care at OSU

DIP- Exclusion Criteria:

* Individuals who cannot tolerate a 2-hour oral glucose tolerance test (OGTT) (i.e. history of gastric bypass)
* Not English or Spanish speaking

PP CARE Inclusion criteria: Enrolled DIP participants who are English speaking will be eligible for PP CARE follow up if they are between 12 and 24 months postpartum.

PP CARE Exclusion criteria: Spanish speaking DIP participants will be excluded because the study team does not include anyone who is Spanish speaking.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is restricted to pregnant individuals.
Enrollment: 104 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of postpartum diabetes mellitus screening | From delivery to up to 12 weeks postpartum
  For patients randomized to inpatient immediate postpartum OGTT, completion of the inpatient test will be confirmed and documented by study staff prior to patient discharge. For patients randomized to the inpatient immediate postpartum OGTT who do not undergo inpatient testing and for patients randomized to the outpatient 4-12 week OGTT, individuals will receive an electronic survey via email at 12 weeks inquiring as to whether they underwent postpartum outpatient OGTT and about the results of testing, if performed.
Patient reported outcome of postpartum Cardiovascular health (CVH) counseling received within the first 12 months after delivery | Within the first 12 months after delivery
  Patient reported outcome of postpartum CVH counseling received within the first 12 months after delivery measured with modified questions from the Pregnancy Risk Assessment Monitoring System (PRAMS) Phase 9 Core Mail Questionnaire and the clinical outcome of postpartum dysglycemia defined as a diagnosis of prediabetes or type 2 diabetes within the first 12 months after delivery.
Patient perspectives, preferences and barriers to engagement with respective to postpartum interventions to improve CVH. | Between 12 and 24 months postpartum
  Semi-structured virtual interviews will be performed including questions that encompass patient perspectives, preferences and barriers to engagement with respective to postpartum interventions to improve CVH.

SECONDARY OUTCOMES:
Risk perception and lifestyle modification | From delivery to up to 12 weeks postpartum
  "What do you think your risk or chance is for getting diabetes over the next 10 years?" (Responses: "almost no chance," "a slight chance," "a moderate chance," or "a high chance.")
  "If you don't change your lifestyle behaviors, such as diet or exercise, what is your risk or chance of getting diabetes over the next 10 years?" (Responses: "almost no chance," "a slight chance," "a moderate chance," or "a high chance.")
  "Have you recently made changes in any lifestyle behaviors that you believe will lower your chance of getting diabetes?" (Responses: yes, no)
  "Are you planning to make changes in any lifestyle behaviors in the near future that you believe will lower your chances of getting diabetes?" (Responses: yes, no)
Rates of primary care provider (PCP) visits within 1 year of delivery | Within 1 year postpartum
  All individuals will be sent an electronic survey via email inquiring as to whether they have attended a visit with a primary care provider (internal medicine, family medicine or primary care nurse practitioner) and for what reason since the time of their delivery.
Risk Perception Survey for Developing Diabetes | From delivery to up to 12 weeks postpartum
  The survey comprises 53 items and has four subscales and other individual items to address various dimensions of risk perception. Risk perception will be assessed as both continuous scales and as a dichotomous outcome ("no chance" and "slight chance" will be categorized as "low" risk perception, and "moderate chance" and "high chance" will be categorized as "high" risk perception.
Diabetes Treatment Satisfaction Questionnaire | From delivery to up to 12 weeks postpartum
  8 question survey will be scored as a continuous scale.
Prediabetes or type 2 diabetes | Within 1 year postpartum
  Prediabetes: OGTT between 140 to 199 mg/dl AND/OR A1c 5.7% to 6.4% AND/OR patient self-report Type 2 diabetes: OGTT 200 mg/dl or higher AND/OR A1c 6.5% or higher AND/OR patient self-report

CONTACTS AND LOCATIONS:
Overall Officials: Christine Field, MD, MPH, Principal Investigator — Ohio State University; Kartik K Venkatesh, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No